CLINICAL TRIAL: NCT05615857
Title: Endocuff Enhanced Colonoscopy: Does it Improve Polyp Detection and Make Rectal Retroflexion Unnecessary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Montfort (Other)
Collaborators: AFP Innovation Fund (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 22-23-04-002
Record Dates: First submitted 2022-10-03; First posted 2022-11-14 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; Colonic Polyps
Keywords: Endocuff; Retroflexion; Colonoscopy; Polyp detection; Screening
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Intervention Model Description: We are to count the number of adenomas and polyps identified per patient while using the Endocuff. These numbers will be compared to the number of identified adenomas and polyps found without the use of the Endocuff retrospectively. In addition, the number of adenomas and polyps found in the rectum while using the Endocuff will be compared to the numbers of adenomas and polyps found with retroflexion without the use of Endocuff. Once the colonoscopy is complete, the patient's level of comfort during the procedure will be documented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Colonoscopy without Endocuff (No Intervention): No Endocuff inserted proximally to colonoscope and use of retroflexion
- Colonoscopy with Endocuff (Experimental): Endocuff inserted proximally to colonoscope, no use of retroflexion
  Interventions: Device: Use of Endocuff during colonoscopy

INTERVENTIONS:
Device: Use of Endocuff during colonoscopy — We will be adding the Endocuff device to the proximal end of the colonoscope, adding an additional tool to facilitate the visualization of the difficult-to-see mucosal areas as well as the rectum. There will be no need for retroflexion to evaluate the colon
  Arms: Colonoscopy with Endocuff

SUMMARY:
The investigators hope that this project will determine if the Endocuff device is a useful adjunct during colonoscopy by optimizing polyp detection and eliminating the need for the painful rectal retroflexion. As such, by improving polyp detection and eliminating the need for rectal retroflexion, it will directly reduce the likelihood of colon cancer and improve patient comfort respectively.

DETAILED DESCRIPTION:
Every day, 73 Canadians are diagnosed with colorectal cancer. This cancer is the third most diagnosed type of cancer in Canada while being the second and third most deadly cancer for men and women respectively. In addition, it accounts for 12% of all cancer diagnoses and cancer deaths for both sexes in 2020. Fortunately, colorectal cancer incidence and mortality rates have been steadily declining in the recent years. This can be attributed to the development of new screening methods and devices assisting in a more reliable identification of polyps as well as removal during colonoscopy. This is essential to prevent cancer as these usually asymptomatic and harmless clusters of atypical cells can turn into cancers, and become fatal if they can progress to a later stage of their development. The Endocuff is a new colonoscopy assisting device designed to aid physicians to maneuver inside the colon, allowing for increased detection of polyps that stay hidden between folds in the colon. By its flexible and hinged arms, the Endocuff is designed to gently flatten the large colonic folds during withdrawal of the colonoscope, bringing the difficult-to-see mucosa to view. The Endocuff also may assist in the view of the rectum, being the last area of the colon and difficult to assess. Usually, a painful procedure called a retroflexion is used to help see this area. However, this pain can limit the evaluation and impact polyp diagnosis in the rectum. In this study, the investigators aspire to answer these following questions: (1) Can the Endocuff improve polyp detection? (2) Can the Endocuff replace the need for retroflexion in the rectum?

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing a colonoscopy during the study period
* Procedure being performed by a gastroenterologist (i.e., surgeons are excluded)

Exclusion Criteria:

* Inflammatory Bowel Disease
* Hereditary Mixed Polyposis Syndrome
* Diverticulitis
* Colonic stricture
* Toxic Megacolon
* Previous Colon surgery, excluding appendectomy
* Radiation therapy to abdomen or pelvis
* Pregnancy/Lactation
* Anticoagulant use
* Suffered stroke or ischemia in previous 3 months
* Being deemed too risky by investigator
* FIT positive
* Poor preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Increase in Polyp Detection Rates when using the Endocuff Enhanced Colonoscopy. | 1 hour
  Comparing Polyp Detection Rate when using the Endocuff Enhanced Colonoscopy to retrospective conventional colonoscopy.
Number of participants endorsing a comfortable procedure when using the Endocuff assisted colonoscopy assessed by Numerical Rating Scale (NRS). | 1 hour
  Results of Numerical Rating Scale pain score when evaluating the rectum with the Endocuff.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Hassard, MD, Principal Investigator — Hopital Montfort; Christine-Nadia Compas, CRC, Study Director — Hopital Montfort
Locations (1):
- Hopital Montfort, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No